CLINICAL TRIAL: NCT07290764
Title: Survival Analysis of Surgical Resection Versus Observation in Patients With Initially Unresectable Hepatocellular Carcinoma Achieving Complete Response After Systemic Therapy: A Multicenter, Real-World Study
Brief Title: Survival Analysis of Surgical Resection Versus Observation in Patients With Initially uHCC Achieving CR After Systemic Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Mao-Lin Yan, professor, Fujian Provincial Hospital
Other Study IDs: TALENP007
Record Dates: First submitted 2025-11-23; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Resection: Patients who with initially unresectable hepatocellular carcinoma achieved complete response after conversion therapy received surgical resection
  Interventions: Procedure: Surgery
- Observation: Patients who with initially unresectable hepatocellular carcinoma achieved complete response after conversion therapy didn't receive surgical resection

INTERVENTIONS:
Procedure: Surgery — Surgical Resection Versus Observation in Patients with Initially Unresectable Hepatocellular Carcinoma Achieving Complete Response After Systemic Therapy
  Groups: Surgical Resection

SUMMARY:
This study aims to further explore the survival benefits of surgical resection after achieving CR in initial uHCC after systemic treatment and the timing of discontinuing systemic treatment

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75
2. Child-Pugh: A/B grade
3. ECOG score: ≤1 point
4. The clinical or pathological diagnosis is consistent with primary HCC, and it has been evaluated by two senior hepatobiliary surgeons as surgically unresectable (including multiple intrahepatic lesions, local vascular invasion, local lymph node metastasis, and distant metastasis).
5. According to the mRECIST criteria, the patient has at least one measurable lesion (the long diameter of the measurable lesion on CT/MRI scans is ≥10mm, and the measurable lesion has not previously received local treatments such as interventional therapy, radiotherapy, or cryotherapy)
6. Patients who achieved CR in tumor response after conversion therapy (based on systemic therapy) (rCR definition: The lesion is completely necrotic as evaluated by enhanced CT/MRI according to the mRECIST criteria；cCR is defined as: reaching rCR according to mRECIST criteria, having no distant metastatic lesions, normal AFP and DCP indicators, and maintaining the above criteria for ≥4weeks); Moreover, it can be surgically removed, with no contraindications for surgery or anesthesia
7. The expected survival time is more than three months
8. The functional indicators of important organs should meet the following requirements: · Blood routine: Absolute neutrophil count ≥ 1.5 × 109/L, Hb ≥ 9.0 g/L, PLT ≥ 75 × 109/L; · Liver function: Total bilirubin ≤ 1.5 times the upper limit of normal value (ULN) (for those with obstructive jaundice, after biliary drainage, it should be ≤ 2.5 times ULN); Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) ≤ 5 times ULN, Albumin ≥ 30 g/L; · Kidney function: Serum creatinine ≤ 1.5 mg/dL, Creatinine clearance rate ≥ 60 ml/min; · Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.
9. No history of severe arrhythmia, heart failure, etc. There is no history of severe ventilation dysfunction or serious pulmonary infection
10. Fertile women should agree to use contraceptive measures during the medication period and for 6 months after the medication is stopped; within 7 days before the study enrollment, the serum or urine pregnancy test must be negative, and the patient must be non-lactating. For male patients, they should agree to use contraceptive measures during the study period and for 6 months after the study is over

Exclusion Criteria:

1. Those who have had other malignant tumor histories within the past 5 years or simultaneously, but have been cured, such as skin basal cell carcinoma, cervical carcinoma in situ, and thyroid papillary carcinoma, are excluded
2. Patients who have received organ transplants in the past or are planning to receive organ transplants
3. Patients with any active autoimmune diseases or those with autoimmune diseases and expected recurrence (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes)
4. Have a history of immune deficiency; Patients who are currently undergoing immunosuppressant or systemic hormone therapy to achieve immunosuppressive effects and are still using them within two weeks prior to signing the informed consent form
5. Known hereditary or acquired bleeding disorders (such as coagulation dysfunction) or thrombosis tendencies, such as in patients with hemophilia; currently using or having used full-dose oral or injectable anticoagulant or thrombolytic drugs for therapeutic purposes (allowing for the preventive use of low-dose aspirin or low-molecular-weight heparin within 10 days prior to the start of the study treatment)
6. Within 4 weeks prior to the first use of the investigational drug, there was a severe infection, such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc.; the baseline chest imaging examination indicated active pulmonary inflammation; within 2 weeks prior to the first use of the investigational drug, there were symptoms and signs of infection or the need for oral or intravenous antibiotic treatment (excluding the use of antibiotics for prophylaxis)
7. Patients with concurrent mental disorders; Has a history of abuse of psychotropic drugs, alcoholism and drug abuse
8. Pregnant or lactating women
9. Those who, as determined by the researchers, are not suitable to participate in this trial for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with initially unresectable hepatocellular carcinoma, the tumor response reached complete remission after systematic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 729 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
three-year OS rate | "From date of enrollment until the date of date of death from any cause, assessed up to 100 months"
  The ratio of the number of survivors from the start of systemic treatment until 3 years to the initial enrollment

SECONDARY OUTCOMES:
progression-free survival | "From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months"
  The period from the initiation of systemic treatment until disease progression, death or loss to follow-up
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 100 months
  The time from the start of systemic treatment until death or loss to follow-up
Treatment-related adverse events | From date of enrollment until the date of death from any cause, assessed up to 100 months
  The incidence rate, occurrence spectrum and severity of adverse events (AE) and serious adverse events (SAE), as well as the outliers of laboratory indicators, were judged according to the NCI-CTCAE V5.0 standard. Dose suspension rate and dose termination rate caused by adverse events

OTHER OUTCOMES:
Time to drug-off | From date of enrollment until the date of drug-off or death from any cause, which come first, assessed up to 100 months
  The time from the initiation of systemic treatment to the assessment of clinical complete response of the tumor and the subsequent discontinuation of systemic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou University Affiliated Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not publicly available due to privacy reasons but are available from the corresponding author upon reasonable request.